CLINICAL TRIAL: NCT06132061
Title: Research on Three-level Prevention and Intervention for Elderly Depression in Urban Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Yunnan University (Other)
Responsible Party: Principal Investigator, Tan Tang, Lecturer, Department of Social Work, Affiliated Hospital of Yunnan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023221
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2023-11

CONDITIONS: Depression in Old Age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group for universal prevention (Experimental): Level 1 intervention (universal prevention) group
  Interventions: Other: universal prevention
- Intervention group for selective prevention (Experimental): Level 2 intervention(selective prevention) group
  Interventions: Other: selective prevention
- Intervention group for targeted prevention (Experimental): Level 3 intervention(targeted prevention) group
  Interventions: Other: targeted prevention
- Control group (Other)
  Interventions: Other: Waiting treatment.

INTERVENTIONS:
Other: universal prevention — Health education related to depression to strengthen the participants' self-care skills to reduce sub-health risk factors.
  Arms: Intervention group for universal prevention
Other: selective prevention — Psychosocial interventions (including but not limited to cognitive behavioral therapy, acceptance commitment therapy, mindfulness training) aimed at risk factors to prevent more severe depressive symptoms.
  Arms: Intervention group for selective prevention
Other: targeted prevention — Therapeutic psychosocial interventions (including but not limited to cognitive behavioral therapy, acceptance commitment therapy, mindfulness training) to reduce patients' depressive symptoms.
  Arms: Intervention group for targeted prevention
Other: Waiting treatment. — Waiting treatment.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to compare the effect of three level interventions(universal prevention, selective prevention and targeted prevention) in elderly depression and find out the most efficient intervention path. The main questions it aims to answer are:

* Whether the pre-disease three-level prevention model (universal prevention, selective prevention and targeted prevention) is applicable for elderly depression in urban communities;
* Which level of intervention has the best effect on elderly depression.

Participants will be given the following treatments:

* Level 1 intervention(universal prevention): Health education related to depression to strengthen the participants' self-care skills to reduce sub-health risk factors.
* Level 2 intervention(selective prevention): Psychosocial interventions (including but not limited to cognitive behavioral therapy, acceptance commitment therapy, mindfulness training) aimed at risk factors to prevent more severe depressive symptoms.
* Level 3 intervention(targeted prevention): Therapeutic psychosocial interventions (including but not limited to cognitive behavioral therapy, acceptance commitment therapy, mindfulness training) to reduce patients' depressive symptoms.

Researchers will compare control group to see if the three levels of intervention have a significant effect.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 and above;
2. Permanent residents of urban communities in China;
3. Geriatric Depression Scale (GDS-15) < 9 points;
4. There are susceptibility factors such as living alone, poverty, and suffering from serious diseases.

Exclusion Criteria:

1. There is suicidal behavior or risk;
2. A history of any other mental illness, including drug or alcohol dependence;
3. Those who have speech and hearing disorder and cannot communicate normally;
4. Geriatric Depression Scale (GDS-15) ≥10 points;
5. Do not agree to participate in the research.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Level of depression | Measurements were taken at baseline, after intervention(3 months after baseline) and 6 months after intervention.The data will be reported through study completion, an average of 1 year.
  A simplified version of Geriatric Depression Scale(GDS-15) will be used to mesure the level of depression. The scale has 15 items and asks the elderly to answer "yes" or "no" based on how they have felt in the past week. The "yes" is 1 point, "no" is 0 points. The higher the score indicates the more obvious depressive symptoms. The total score is 15 points. 0-4 points indicate no depression, 5-9 points indicate mild depression, and 10-15 points indicate moderate to severe depression.

SECONDARY OUTCOMES:
Psychological flexibility | Measurements were taken at baseline, after intervention(3 months after baseline) and 6 months after intervention.The data will be reported through study completion, an average of 1 year.
  Psychological flexibility refers to an individual's ability to be open and flexible to his or her own experiences, thoughts or feelings, which can prompt him or her to take action or make changes when engaged in difficult events. Psychological flexibility can be measured by the simplified Multidimensional Psychological Flexibility Inventory(MPFI-24). The scale consists of 24 items and is divided into two subscales: psychological flexibility (PF) and psychological inflexibility (PI). Each items is rated by the subject on a 6-point Likert scale (1＝never to 6＝always). Higher subscale scores were associated with higher levels of psychological flexibility or psychological inflexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Street, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No